CLINICAL TRIAL: NCT06038162
Title: Evaluation of Integrated Versus Parallel Continuous Renal Replacement Therapy Connection in ECMO Patients: a Randomized Controlled Trial
Brief Title: Evaluation of Integrated Versus Parallel Connection for Renal Replacement Therapy in ECMO Patients
Acronym: EPIC-ECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL22_0894
Record Dates: First submitted 2023-08-31; First posted 2023-09-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Venoarterial Extracorporeal Membrane Oxygenation; Renal Replacement Therapy; Acute Kidney Injury
Keywords: VA-ECMO; RRT; connection; integrated; parallel; hemofilter
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA-ECMO patients with parallel connection (Active Comparator): Patients undergoing VA ECMO with indication for concomitant RRT, assigned to parallel connection group.
  Interventions: Procedure: Parallel connection
- VA-ECMO patients with integrated connection (Active Comparator): Patients undergoing VA ECMO with indication for concomitant RRT, assigned to integrated connection group.
  Interventions: Procedure: Integrated connection

INTERVENTIONS:
Procedure: Parallel connection — The RRT machine is connected on a separate vascular access (dialysis catheter).
  Arms: VA-ECMO patients with parallel connection
Procedure: Integrated connection — A connection of the RRT machine with the input and output lines directly on the ECMO circuit.
  Arms: VA-ECMO patients with integrated connection

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is an extra-corporeal assistance used in case of respiratory or circulatory failure. In case of circulatory failure, ECMO is in the veno-arterial configuration (VA-ECMO). VA-ECMO patients are at high risk of developing acute kidney injury (AKI) and renal replacement therapy (RRT) may be needed in 50% of ECMO patients. Although the administration of RRT in ECMO patients has major implications, no specific recommendations are currently available. The 2020 Kidney Disease: Improving Global Outcomes (KDIGO) international conference identified the evaluation of RRT in these ECMO patients as a research priority.

In 2023, the two main configurations used to administer RRT in ECMO patients are an independent delivery on a separate vascular access (parallel connection) or an integration of the RRT machine directly into the ECMO circuit (integrated connection). The integrated connection may reduce infectious and bleeding complications associated with the use of a second vascular access. However, it can expose the hemofilter and circuit to excessive positive pressures that can trigger pressure alarms in the RRT machine and expose the patient to a theoretical risk of air embolism or hemolysis. Furthermore, there is currently no robust data comparing the hemofilter lifespan with the parallel or with the integrated connection, although the filter lifespan is a crucial parameter to assess the quality of the RRT delivery in the ICU. The investigators recently performed a survey of practices in this context of ECMO patients. The investigators found that both strategies (parallel and integrated connection) are widely used and can be seen as common patient care.

The hypothesis tested in this study is the following: when RRT is integrated to the ECMO circuit, the hemofilter lifespan is non inferior to the one when RRT is delivered on a separate vascular access. Only VA-ECMO patients will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years
* Patient on VA-ECMO who requires the initiation of continuous RRT during VA-ECMO treatment
* Patient with a foreseeable length of stay in intensive care greater than 24 hours

Exclusion Criteria:

* Patient who does not have a vascular capital allowing for the insertion of a new dialysis catheter to administer RRT and therefore cannot be randomized to the parallel connection group
* High pressures monitored on ECMO not allowing direct RRT catherter on ECMO
* Pregnant, parturient, or breastfeeding women
* Patient deprived of liberty by a judicial or administrative decision
* Patient under psychiatric care
* Patient subject to a legal protection measure (guardianship, curators)
* Patient not affiliated to a social security system
* Patient participating in another interventional research study in the field of extra purification renal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2028-02-07 (Estimated); Study Completion 2028-04-07 (Estimated)

PRIMARY OUTCOMES:
Hemofilter change rate | Duration of RRT associated with VA-ECMO up to 60 days
  To assess whether integrated RRT connection in VA-ECMO patients results in a non-inferior hemofilter change rate compared to the parallel connection.
  The hemofilter change rate is defined as the number of hemofilter replacements observed during the period between the start and the end of the RRT session, normalized by the duration of the session.

SECONDARY OUTCOMES:
Proportion of early hemofilter thromboses | Duration of RRT associated with VA-ECMO up to 60 days
  To assess if the integrated RRT connection is associated with a lower proportion of early hemofilter thromboses compared to the parallel connection: number of early hemofilter thromboses normalized by the number of hemofilters used. "Early" is defined as < 24 hours of use.
Proportion of hemofilter thromboses | Duration of RRT associated with VA-ECMO up to 60 days
  To assess if the integrated RRT connection is associated with a lower proportion of hemofilter thromboses compared to the parallel connection: number of hemofilter thromboses normalized by the number of hemofilters used.
Down-time | Duration of RRT associated with VA-ECMO up to 60 days
  To compare the integrated RRT connection to the parallel connection in terms of duration of non-purification periods in relation to the total duration RRT.
Renal function according to KDIGO stage | At hospital discharge up to 60 days after admission
  To assess renal function at hospital discharge or at day 60 after admission.
Number of infectious complications | Duration of RRT associated with VA-ECMO up to 60 days
  To assess whether the integrated RRT connection reduces the number of infectious complications associated with the use of an additional vascular access.
  The infection will be defined as catheter-related in case of documented bacteraemia with positive blood cultures with differential time to positivity or positive catheter culture with the same microorganism.
Number of bleeding complications | Duration of RRT associated with VA-ECMO up to 60 days
  To assess whether the integrated RRT connection reduces bleeding complications associated with the use of an additional vascular access.
  The occurrence of a bleeding syndrome is defined as a bleeding requiring transfusion with collection of the number of red blood cells transfused or requiring an invasive procedure (surgery, embolization), and defined or not as related to dialysis catheter placement or RRT connection to VA-ECMO.
Proportion of ECMO circuit thromboses | Duration of RRT associated with VA-ECMO up to 60 days
  To assess whether the integrated RRT connection does not expose the ECMO circuit to a higher probability of thrombosis The occurrence of thrombosis on the ECMO circuit is defined as a thrombus on any part of the ECMO circuit requiring a change in the circuit or oxygenator, or on the oxygenator resulting in a deleterious effect on oxygenation, or resulting in significant fibrinolysis
Number of hemolysis | Duration of RRT associated with VA-ECMO up to 60 days
  To assess whether the integrated RRT connection does not expose to a higher probability of hemolysis.
  The occurrence of intravascular hemolysis is defined as the occurrence of significant hemolytic anemia.
Number of air embolism | Duration of RRT associated with VA-ECMO up to 60 days
  To assess whether the integrated RRT connection does not expose the patient to a higher probability of air embolism.
  The occurrence of an air embolism is defined as an embolic event with clinical impact of any kind, This occurence is related or not to the use of the dialysis catheter or the connection of the RRT to the VA-ECMO circuit.
Number of days spent in intensive care unit | Duration of RRT associated with VA-ECMO up to 60 days
  To assess whether the integrated RRT connection modifies the intensive care unit length of stay
Death | At 30 days
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Frank BIDAR, MD, Study Chair — Hospices Civils de Lyon
Locations (12):
- France (12):
  - CHU de Bordeaux, GH Sud, Service d'anesthésie-réanimation cardiovasculaire, Hôpital cardiologique, Bordeaux
  - CHU de Clermont Ferrand, Pôle de médecine péri-opératoire/Chirurgie cardiaque, Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalo Universitaire de Dijon, Unité Réanimation Cardio-Vasculaire,, Dijon
  - CHU de Grenoble, Service de réanimation cardiovasculaire et thoracique, Pôle anesthésie réanimation, Hôpital Nord, Grenoble
  - Centre Hospitalo Universitaire de Lille, Institut Coeur Poumon, Lille
  - Hospices Civils de Lyon, Service d'Anesthésie-Réanimation cardiovasculaire, Hôpital Louis Pradel, Lyon
  - CHU de Montpellier, Département d'anesthésie-réanimation, Pôle Cœur-poumons, Hôpital Arnaud de Villeneuve, Montpellier
  - APHP, Institut de Cardiologie, Service d'anesthésie-réanimation cardiovasculaire, Hôpital de la Pitié-Salpêtrière, Paris
  - APHP, Institut de cardiologie, Service de Médecine Intensive Réanimation, Hôpital Pitié-Salpêtrière, Paris
  - CHU de Saint Etienne, Hôpital Bellevue, Service de Réanimation polyvalente et soins intensifs post-opératoires, Saint-Etienne
  - Centre Hospitalo Universitaire de Toulouse, Hôpital Rangueil - Réanimation polyvalente, Toulouse
  - Centre Hospitalo Universitaire de Toulouse, Unité de Chirurgie Cardiaque, Toulouse